CLINICAL TRIAL: NCT04821570
Title: Cancer Therapy and Immunogenicity of COVID Vaccine (CANINE Trial)
Brief Title: To Assess Immunogenicity of Coronavirus Disease 2019 (COVID-19) Vaccine in Cancer Patients Receiving Cancer Treatment
Acronym: CANINE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2021-CANINE
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Lung Cancer; Melanoma (Skin)
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Melanoma | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Chemotherapy (IV and oral)
  Interventions: Biological: COVID-19 Vaccine
- Immunotherapy
  Interventions: Biological: COVID-19 Vaccine
- Chemotherapy + Immunotherapy
  Interventions: Biological: COVID-19 Vaccine
- Cyclin- dependent kinase (CDK) 4/6 inhibitors
  Interventions: Biological: COVID-19 Vaccine
- Stem Cell Transplant recipients
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — Per recommended dosing schedule

SUMMARY:
This is a trial of prospective collection of serial blood samples after administration of COVID-19 vaccine in patients with cancer who are receiving active cancer treatment, planned to start therapy with 14 days of consent, or have had stem cell transplant. Cancer treatments and administration of vaccine are not controlled by the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Males and females age ≥ 18 years
* Patients with breast cancer, lung cancer, malignant melanoma or who have undergone stem cell transplant or chimeric antigen receptor (CAR) T cell therapy for a hematologic malignancy.

Other cancer types including hematologic malignancies may be allowed if they are receiving treatments outlined in section 4.1.4

* Solid Tumor patients and those with hematologic malignancies: Currently receiving active anti-cancer therapy, or planned to start within 14 days, with intravenous cytotoxic chemotherapy (oral or intravenous), intravenous chemoimmunotherapy combination, immunotherapy alone, an oral CDK 4/6 inhibitor. (This does not apply to recipients of stem cell transplant and CAR T therapy)
* Therapy may be neo/adjuvant or for metastatic disease
* Eastern Cooperation Oncology Group (ECOG) Performance status (PS) of 0-2

Exclusion Criteria:

* Life expectancy of < 12 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants undergoing treatment for breast cancer, lung cancer and melanoma with chemotherapy, immunotherapy and/or oral anticancer agents, or have undergone stem cell transplantation
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-03-28 (Estimated); Study Completion 2025-03-28 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) with corresponding 95%confidence interval (CI) at each time point of the entire population and individually of all cohorts | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Pfizer: Baseline, Day 21, Day 51, Day 111, Day 201.
  Elecsys Anti severe acute respiratory syndrome (SARS) coronavirus 2 (CoV 2) S quantitative assay
Geometric mean titer (GMT) with corresponding 95% CI at each time point of the entire population and individually of all cohorts | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Moderna: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 S quantitative assay
Geometric mean titer (GMT) with corresponding 95% CI at each time point of the entire population and individually of all cohorts | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Johnson & Johnson: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 S quantitative assay
Geometric mean fold rise (GMFR) with corresponding 95% CI at each post-baseline timepoint over preinjection baseline | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Moderna: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 S quantitative assay
Geometric mean fold rise (GMFR) with corresponding 95% CI at each post-baseline timepoint over preinjection baseline | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Pfizer baseline, Day 21, Day 51, Day 111, Day 201
  Elecsys Anti SARS CoV 2 S quantitative assay
Geometric mean fold rise (GMFR) with corresponding 95% CI at each post-baseline timepoint over preinjection baseline | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Johnson & Johnson: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 S quantitative assay

SECONDARY OUTCOMES:
Geometric median, minimum and maximum assay titer values for each cohort | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Moderna: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 S quantitative assay
Geometric median, minimum and maximum assay titer values for each cohort | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Pfizer: Baseline, Day 21, Day 51, Day 111, Day 201
  Elecsys Anti SARS CoV 2 S quantitative assay
Geometric median, minimum and maximum assay titer values for each cohort | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Johnson & Johnson: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 S quantitative assay
The number of subjects with fold-rise ≥ 2 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Moderna: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The percentage of subjects with fold-rise ≥ 2 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Moderna: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The number of subjects with fold-rise ≥ 3 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Moderna: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The percentage of subjects with fold-rise ≥ 3 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Moderna: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The number of subjects with fold-rise ≥ 4 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Moderna: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The percentage of subjects with fold-rise ≥ 4 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Moderna: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The number of subjects with fold-rise ≥ 2 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Pfizer: Baseline, Day 21, Day 51, Day 111, Day 201
  Elecsys Anti SARS CoV 2 quantitative assay
The percentage of subjects with fold-rise ≥ 2 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Pfizer: Baseline, Day 21, Day 51, Day 111, Day 201
  Elecsys Anti SARS CoV 2 quantitative assay
The number of subjects with fold-rise ≥ 3 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Pfizer: Baseline, Day 21, Day 51, Day 111, Day 201
  Elecsys Anti SARS CoV 2 quantitative assay
The percentage of subjects with fold-rise ≥ 3 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Pfizer: Baseline, Day 21, Day 51, Day 111, Day 201
  Elecsys Anti SARS CoV 2 quantitative assay
The number of subjects with fold-rise ≥ 4 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Pfizer: Baseline, Day 21, Day 51, Day 111, Day 201
  Elecsys Anti SARS CoV 2 quantitative assay
The percentage of subjects with fold-rise ≥ 4 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Pfizer: Baseline, Day 21, Day 51, Day 111, Day 201
  Elecsys Anti SARS CoV 2 quantitative assay
The number of subjects with fold-rise ≥ 2 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Johnson & Johnson: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The percentage of subjects with fold-rise ≥ 2 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Johnson & Johnson: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The number of subjects with fold-rise ≥ 3 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Johnson & Johnson: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The percentage of subjects with fold-rise ≥ 3 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Johnson & Johnson: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The number of subjects with fold-rise ≥ 4 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Johnson & Johnson: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay
The percentage of subjects with fold-rise ≥ 4 from baseline at each post injection time points with 95% CIs | Participants will have scheduled blood sampling (for immunogenicity assessment) at: For Johnson & Johnson: Baseline, Day 29, Day 57, Day 119, Day 209
  Elecsys Anti SARS CoV 2 quantitative assay

CONTACTS AND LOCATIONS:
Overall Officials: Qamar Khan, MD, Principal Investigator — University of Kansas
Locations (1):
- The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided